CLINICAL TRIAL: NCT05996172
Title: Swift Outpatient Alternatives for Rapid Stabilization
Acronym: SOARS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Molly Adrian, Associate Professor, Psychiatry and Behavioral Sciences, University of Washington
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00016898; P50MH129708 (NIH)
Record Dates: First submitted 2023-06-19; First posted 2023-08-18 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Suicidal Ideation; Suicide Attempt
MeSH Terms: conditions — Suicidal Ideation; Suicide, Attempted

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- CAMS Single Session Consultation (SSC) (Active Comparator): CAMS is a clinical intervention designed to modify how clinicians engage, assess and plan treatment with suicidal patients. The foundational brief intervention that all participants will receive includes 1 90-minute session of CAMS assessment and planning interview with follow-up care navigation.
  Interventions: Behavioral: CAMS Single Session Consultation
- CAMS SSC + Driver-Focused Skills Training (Active Comparator): Specific skills are taught to youth based on CAMS drivers/case conceptualization of suicidality. Based on our pilot work, the common components of treatment include explicit coaching in skills informed by evidence-based treatments like Dialectical Behavior Therapy (DBT), Cognitive Behavioral Therapy (CBT), and Behavioral Activation (BA). Skills are drawn from the following 3 domains: emotion regulation and crisis survival skills (e.g., paced breathing, use of temperature and exercise to alter mood, Hope Box), behavioral activation strategies (e.g., goal-directed behavior, scheduling of activities, problem-solving) and communication skills (communication around suicidality, validation of self and others, making clear requests/DEAR MAN). Youth assigned to the Ongoing CAMS Intervention condition will receive three, 50-minute sessions that include the interim SSF and driver focused treatment encompassing skills instruction, in-session practice, and assigned homework.
  Interventions: Behavioral: CAMS Single Session Consultation; Behavioral: Driver Focused Skills Training
- CAMS SSC + Caregiver Skills Building (Active Comparator): Caregivers will receive 3, 30-minute modules across 3 sessions that provide explicit coaching in several skills. Module content will include 1) psychoeducation on suicidality and the escalation cycle and creation of a communication plan related to responding to youth suicidality (i.e., Crisis Escalation and Communication Plan); 2) positive communication and relationship building strategies including reflective listening, validation, and how to implement regular teen-directed one-on-one time; and 3) setting up behavioral expectations, house rules, and using positive reinforcement based contingency management in the home (i.e., targeted praise, using rewards to promote more effective behaviors). All modules will include didactic skill building, role-play of skill use with the therapist, and a check-in with the youth and youth therapist to collaboratively problem-solve barriers to use of skills.
  Interventions: Behavioral: CAMS Single Session Consultation; Behavioral: Caregiver Skills Training
- CAMS SSC + Lethal Means Safety (Active Comparator): The CAMS Therapeutic Assessment incorporates low levels of lethal means restriction (see above). Experimental Intervention Component 4 will provide a high level of lethal means restriction that includes the evaluation of the need for a lock box, the provision of a lock box if needed, structured process for evaluating home safety in each room of the house, specific directives to accomplish, follow up with the clinician, and problem-solving barriers to lethal means restriction over two, 30-minute modules delivered across 2 sessions.
  Interventions: Behavioral: CAMS Single Session Consultation; Behavioral: Lethal Means Safety
- CAMS SSC + Driver Focused Skills Training + Caregiver training (Active Comparator): This arm includes CAMS SSC, 3 sessions of youth facing driver focused skills, and 3 sessions of caregiver skills training.
  Interventions: Behavioral: CAMS Single Session Consultation; Behavioral: Driver Focused Skills Training; Behavioral: Caregiver Skills Training
- CAMS SSC + Driver Focused Skills Training + Lethal Means Safety (Active Comparator): This arm includes the CAMS single session intervention, 3 sessions of skills training for the youth, and lethal means safety for caregiver.
  Interventions: Behavioral: CAMS Single Session Consultation; Behavioral: Driver Focused Skills Training; Behavioral: Lethal Means Safety
- CAMS SSC + Caregiver Skills Training + Lethal Mean Safety (Active Comparator): The arm includes the CAMS single session intervention, 3 sessions caregiver skills training and lethal means safety.
  Interventions: Behavioral: CAMS Single Session Consultation; Behavioral: Caregiver Skills Training; Behavioral: Lethal Means Safety
- CAMS SSC + Driver Focused Skills Training + Caregiver Skills + Lethal Means Safety (Active Comparator): This arm includes the single session intervention, youth skills training, caregiver skills training and lethal means safety.
  Interventions: Behavioral: CAMS Single Session Consultation; Behavioral: Driver Focused Skills Training; Behavioral: Caregiver Skills Training; Behavioral: Lethal Means Safety

INTERVENTIONS:
Behavioral: CAMS Single Session Consultation — CAMS is a clinical intervention designed to modify how clinicians engage, assess and plan treatment with suicidal patients. The foundational brief intervention that all participants will receive includes 1 90-minute session of CAMS assessment and planning interview with follow-up care navigation. CAMS is based around a model of STB which states that youth become suicidal in response to overwhelming pain, and treatment identifies and targets the drivers of suicide as the primary focus of assessment and intervention.
Behavioral: Driver Focused Skills Training — The CAMS approach focuses on therapeutic assessment, collaborative identification and treatment of the patient-defined STB drivers (i.e., the problems that make suicide compelling to the patient) and utilizes problem-focused treatment sessions to address the drivers in order to reduce the wish to die. In the SOARS brief intervention model, specific skills are taught to youth based on CAMS drivers/case conceptualization of suicidality.
  Arms: CAMS SSC + Driver Focused Skills Training + Caregiver Skills + Lethal Means Safety; CAMS SSC + Driver Focused Skills Training + Caregiver training; CAMS SSC + Driver Focused Skills Training + Lethal Means Safety; CAMS SSC + Driver-Focused Skills Training
Behavioral: Caregiver Skills Training — Caregivers will receive 3, 30-minute modules across 3 sessions that provide explicit coaching in several skills adapted from evidence-based treatments for youth suicidality including DBT and CBT.48,49 Module content will include 1) psychoeducation on suicidality and the escalation cycle and creation of a communication plan related to responding to youth suicidality (i.e., Crisis Escalation and Communication Plan); 2) positive communication and relationship building strategies including reflective listening, validation, and how to implement regular teen-directed one-on-one time; and 3) setting up behavioral expectations, house rules, and using positive reinforcement based contingency management in the home (i.e., targeted praise, using rewards to promote more effective behaviors). All modules will include didactic skill building, role-play of skill use with the therapist, and a check-in with the youth and youth therapist to collaboratively problem-solve barriers to use of skills.
  Arms: CAMS SSC + Caregiver Skills Building; CAMS SSC + Caregiver Skills Training + Lethal Mean Safety; CAMS SSC + Driver Focused Skills Training + Caregiver Skills + Lethal Means Safety; CAMS SSC + Driver Focused Skills Training + Caregiver training
Behavioral: Lethal Means Safety — The CAMS Therapeutic Assessment incorporates low levels of lethal means restriction (see above). Experimental Intervention Component 4 will provide a high level of lethal means restriction that includes the evaluation of the need for a lock box, the provision of a lock box if needed, structured process for evaluating home safety in each room of the house, specific directives to accomplish, follow up with the clinician, and problem-solving barriers to lethal means safety over two, 30-minute modules delivered across 2 sessions.
  Arms: CAMS SSC + Caregiver Skills Training + Lethal Mean Safety; CAMS SSC + Driver Focused Skills Training + Caregiver Skills + Lethal Means Safety; CAMS SSC + Driver Focused Skills Training + Lethal Means Safety; CAMS SSC + Lethal Means Safety

SUMMARY:
The goal of this clinical trial is to improve the effective outpatient management of acute youth suicide risk by optimizing intervention components to build an efficient, evidence-based intervention that is responsive to the needs of, and coordinated with, providers in primary care settings. The main questions are:

1. What is the strongest combination of SOARS components associated with reduction in youth suicidal thoughts and behavior (STB)?
2. Do age and STB history moderate the impact of the effects of the SOARS intervention components?
3. Do therapeutic alliance, youth and caregiver self-efficacy account for changes in youth STBs?
4. What helps medical outpatient providers refer to SOARS and continue care after SOARS?

DETAILED DESCRIPTION:
The investigators are comparing different treatment sequences for suicidal thoughts and behaviors. The treatment package families are assigned will be determined by randomization.

All participants will receive 1 session of Collaborative Assessment and Management of Suicidality (CAMS) and care management. CAMS treatment primarily focuses on working with a therapist to understand the reasons why the participants are thinking about suicide Additional components which the participant may be randomly assigned to receive include coping skills training for youth, skills training for parents, and additional safety strategies. Each treatment type is designed to help adolescents and young adults with suicide risk.

Participants will be randomly assigned to an intervention sequence for a minimum of 1 session (120 minutes) and maximum of 8 sessions (440 minutes, divided across separate youth and caregiver components).

Caregivers will receive at least 1 session and a maximum of 4 sessions. Depending on the randomization, caregivers may be assigned to receive skills related to caregiving and safe storage of items that could be used for harm.

To see how the treatment is going participants will receive study assessments at the beginning of the study, 1-month, and 2-months. Study assessments will ask about demographics, suicide attempts, suicidal ideation, non-suicidal self-injury, experiences with treatment, substance use, and social experiences. The research team will also collect information from medical records.

ELIGIBILITY:
Inclusion Criteria:

* Acute suicidal thoughts or past month suicide attempt as reported on positive responses to the Ask Suicide Screening Questionnaire (ASQ),

Exclusion Criteria:

* urgent medical care secondary to self-injurious behavior, psychosis, eating disorder that requires full or partial inpatient care, or
* intellectual disability warranting a different treatment pathway;
* limited English, Spanish, Vietnamese, or Chinese proficiency that would interfere with ability to complete study assessments;
* unwillingness to participate in psychotherapy,
* caregiver unwilling or ineligible to participate;
* and previous enrollment in SOARS program or other P50 project as to not confuse longitudinal follow-up.

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 184 (Estimated)
Dates: Start 2023-11-09 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Harkavy-Asnis Suicide Scale | baseline, 1, and 2 month follow up
  This measure assesses the frequency of suicidal ideation on a 5-point Likert scale, with 0 indicating "never" and 4 indicating "most or all of the time". Higher scores reflect higher severity and frequency of suicidal ideation.

SECONDARY OUTCOMES:
Columbia Suicide Severity Rating Scale (C-SSRS) | baseline, 1, & 2 month follow up
  ASuicidal thoughts and behaviors. Suicide ideation is rated on a scale of 1 to 5, with higher numbers reflecting more severe ideation. Suicidal behaviors are count measures, with higher numbers reflecting more attempts.

CONTACTS AND LOCATIONS:
Overall Officials: Molly Adrian, Ph.D., Principal Investigator — University of Washington
Locations (1):
- Seattle Children's, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No